CLINICAL TRIAL: NCT05867420
Title: A Phase 1 Dose Escalation Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of ASKG915 in Patients With Selected Advanced Solid Tumors
Brief Title: A Study of ASKG915 in Patients With Selected Advanced Solid Tumors.
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: AskGene Pharma, Inc. (Industry)
Collaborators: Jiangsu Aosaikang Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ASKG915-101
Record Dates: First submitted 2023-05-04; First posted 2023-05-22 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Advanced Solid Tumors
Keywords: PD-1/IL-15
MeSH Terms: interventions — Paclitaxel; Bevacizumab; HMPL-013; Docetaxel

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- ASKG915 (Experimental): For monotherapy (Part A and Part B), subjects will receive ASKG915 via intravenous (IV) infusion at a frequency of once every 3 weeks (Q3W) or once every 4 weeks (Q4W), at either the prespecified dose levels or the levels determined by the Study Review Committee (SRC).
  Interventions: Biological: ASKG915
- ASKG915 combination with SOC (Experimental): For combination therapy phase (Part C), subjects will receive ASKG915 at recommended dose levels via intravenous (IV) infusion, administered once every 3 weeks (Q3W) or once every 4 weeks (Q4W), and in combination with the standard treatment regimen for the selected tumor types.
  Interventions: Biological: ASKG915; Drug: Paclitaxel + Bevacizumab; Drug: Fruquintinib; Drug: Docetaxel

INTERVENTIONS:
Biological: ASKG915 — ASKG915 is administered intravenously at a scheduled dose. The drug was given once every 3 weeks or 4 weeks for a cycle.
Drug: Paclitaxel + Bevacizumab — Paclitaxel is administered intravenously at a dose of 80 mg/m², once weekly on a 21-day cycle.
  Bevacizumab is administered intravenously at dose of 15mg/kg, once every 3 weeks on a 21-day cycle.
  Arms: ASKG915 combination with SOC
Drug: Fruquintinib — The recommended dose of Fruquintinib is 5 mg orally once daily, with or without food for the first 21 days of each 28-day cycle.
  Arms: ASKG915 combination with SOC
Drug: Docetaxel — Docetaxel is administered intravenously at 75 mg/m², once every 3 weeks on a 21-day cycle.
  Arms: ASKG915 combination with SOC

SUMMARY:
The study is a dose-escalation and dose-expansion study to evaluate the safety, tolerability, and pharmacokinetics of ASKG915 as a single agent or in combination with standard of care (SOC) in patients with selected types of advanced solid tumors.

DETAILED DESCRIPTION:
Monotherapy:

A dose-escalation (Part A) and expansion (Part B) study of ASKG915 monotherapy was initiated to evaluate the safety, tolerability, pharmacokinetics (PK), and pharmacodynamics (PD) in patients with advanced solid tumors.

Combination therapy:

A dose-optimization (Part C) srudy of ASKG915 in combination with standard of care (SOC) in patients was conducted to evaluate the safety, tolerability, pharmacokinetics (PK), and pharmacodynamics (PD) in patients with selected types of advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed advanced malignant tumor that is refractory to or intolerant of all standard therapy or for which no standard therapy is available.
2. ECOG performance status of ≤ 2.
3. Life expectancy of ≥ 3 months.
4. The results of the laboratory tests must meet all criteria.

Exclusion Criteria:

1. Patients have received antitumor therapy during the first 4 weeks before study drug use.
2. Received a live attenuated vaccine within 4 weeks prior to C1D1.
3. Known cerebral parenchymal metastasis or meningeal metastasis.
4. History of serious cardiovascular or cerebrovascular diseases.
5. Active or recurrent autoimmune diseases.
6. History of ascites or pleural effusion requiring drainage.
7. Pregnant or lactating or planning to become pregnant at any time during the study, including the Follow-up Period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 594 (Estimated)
Dates: Start 2023-08-02 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Dose limiting toxicities (DLTs) | 21days or 28 days
  To evaluate the safery of ASKG915 in subjects.
Adverse events(AEs) | From the first dose to 30 days after the last dose
  To evaluate the safery of ASKG915 in subjects.

SECONDARY OUTCOMES:
Maximum plasma concentration (Cmax) | Until treatment discontinuation or for a maximum of 2 years
  To evaluate the systemic pharmacokinetics of ASKG915 in subjects.
Area under the concentration time curve (AUC) | Until treatment discontinuation or for a maximum of 2 years
  To evaluate the systemic pharmacokinetics of ASKG915 in subjects.
Plasma clearance rate (CL) | Until treatment discontinuation or for a maximum of 2 years
  To evaluate the systemic pharmacokinetics of ASKG915 in subjects.
Evaluation of immunogenicity | Until treatment discontinuation or for a maximum of 2 years
  Incidence of anti-drug antibodies (ADA)
Objective Response Rate (ORR) | Until disease progression or for a maximum of 2 years
  The percentage of patients having a best overall response of complete response (CR) or partial response (PR)
Duration of response (DOR) | Until disease progression or for a maximum of 2 years
  The DOR will be calculated from the time of initial response (PR or better that is subsequently confirmed) to progression (after PR) or death
Progression-free survival (PFS) | Until disease progression or for a maximum of 2 years
  PFS is defined as the time from the date of first dose of study treatment until the date of progressive disease or death, whichever is earlier

CONTACTS AND LOCATIONS:
Overall Officials: Jing Chen, MD, Study Director — Ask-Gene Pharma, Inc.
Locations (4):
- United States (2):
  - Columbia University Irving Medical Center, New York, New York
  - UPMC Hillman Cancer Center, Pittsburgh, Pennsylvania
- China (2):
  - Peking University Cancer Hospital, Beijing, Beijing Municipality
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality